CLINICAL TRIAL: NCT01752010
Title: A Randomized Study Comparing the Tennant BioModulator to Transcutaneous Electrical Nerve Stimulation (TENS) and Traditional Chinese Acupuncture for the Symptomatic Treatment of Chronic Pain Among Injured Service Members.
Brief Title: Comparing Acupuncture, BioModulator, and Transcutaneous Electrical Nerve Stimulation for Symptomatic Treatment of Chronic Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samueli Institute for Information Biology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2009.098
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Pain; Depression; PTSD Symptoms; Sleep
MeSH Terms: conditions — Chronic Pain; Depression | interventions — Transcutaneous Electric Nerve Stimulation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acupuncture Treatment (Active Comparator): Traditional Chinese acupuncture.
  Interventions: Other: Traditional Chinese Acupuncture
- Tennant™ Biomodulator Treatment (Active Comparator)
  Interventions: Device: Tennant™ Biomodulator Treatment
- Transcutaneous electrical nerve stimulation (TENS) Treatment (Active Comparator)
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS) Treatment

INTERVENTIONS:
Other: Traditional Chinese Acupuncture — Treatment will be performed by an experienced provider, and may include insertion of sterile 32-gage (0.25mm) acupuncture needles on any part of the body that can be needled while the subject is lying prone with their head in a face cradle. The needles are usually retained for 20-30 minutes along various meridian points identified by the practitioner as being "blocked." Needles will be inserted to the depth typically recommended for the particular point of concern; generally 1 to 3cm. There are no constraints on the number of needles used. Acupuncture points are points of lower resistance and higher electrical conductance than the surrounding tissue. Placing the acupuncture needles into points identified as blocked is believed to help restore the flow of energy and stimulates the release of endorphins. The subject's level of pain is assessed on a 0-10 pain scale. Thirty minute acupuncture treatments will be given by the provider once a week for 6 weeks at the pain clinic.
  Arms: Acupuncture Treatment
Device: Tennant™ Biomodulator Treatment — An FDA-approved Tennant™ 650 BioModulator will be used to deliver electrical stimulation. The device will be applied directly on top of the subject's area of pain for one minute; power is adjusted until the subject feels a slight tingle. Random variations of pulse amplitude are set from zero to a chosen comfort limit. A feedback mechanism is provided by the constant monitoring of skin impedance. The device is then pressed onto the site of pain and rotated counter-clockwise. After a minute, the device is placed on the opposite side of the pain site and the procedure repeated. The subject's level of pain is assessed on a 0-10 pain scale. At no time is the level of electrical stimulation allowed to cause sustained pain. The subject will receive a weekly 15 minute visit that includes a treatment provided by the pain provider. The provider will teach the subject how to use the machine by themselves and instruct the subject to use the machine twice a day on their own during the study.
  Arms: Tennant™ Biomodulator Treatment
Device: Transcutaneous electrical nerve stimulation (TENS) Treatment — An FDA-approved Empi™ TENS unit will be used to deliver the transcutaneous electrical nerve stimulation. The low frequency TENS unit will be applied to the subject's area of pain by the use of four integrated self-adhering 5x5 cm electrodes. The electrodes will be positioned at a distance of 3 cm and centered over the area that is most painful. The device rapidly delivers therapeutic electrical currents at various frequencies off and on 150 times a second. The subject's level of pain is assessed on a 0-10 pain scale. At no time is the level of electrical stimulation allowed to cause sustained pain. The subject will receive a weekly 15 minute visit that includes a treatment provided by the pain provider. The provider will teach the subject how to use the machine by themselves and instruct the subject to use the machine twice a day on their own during the study.
  Arms: Transcutaneous electrical nerve stimulation (TENS) Treatment

SUMMARY:
The primary objective of this preliminary study is to compare the Tennant BioModulator with Transcutaneous Electrical Nerve Stimulation (TENS) and Traditional Chinese Acupuncture for the management of chronic pain among injured service members. The secondary objective is to investigate any associative effects or benefits on sleep, Post-Traumatic Stress Disorder (PTSD) symptoms, or depression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be Injured service members between the ages of 18 and 60, inclusive;
* The pain must have been present for 3 months or greater prior to entry into the study;
* Subjects must agree to follow the medication regime as directed by the pain clinic provider for the duration of the study;
* Subjects must be able to speak and read English and understand study procedures

Exclusion Criteria:

* Epilepsy
* Pregnancy, or considering pregnancy within the study time-frame
* Pacemaker
* History of cardiac arrhythmias
* Implantable devices (AICD, pump, etc.)
* Surgical intervention during the past month for the treatment of low back pain or its underlying etiology
* Documented history of prescription medication abuse
* Abuse of illicit drugs within the last 6 months
* Participation in a clinical trial for an investigational drug and/or agent within 30 days prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2010-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Chronic pain | Baseline; post-intervention; one-month follow up.

SECONDARY OUTCOMES:
Depression, PTSD symptoms, Sleep. | Baseline; post-intervention; one-month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schlicher, PhD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

REFERENCES:
- [Derived] Peacock KS, Stoerkel E, Libretto S, Zhang W, Inman A, Schlicher M, Cowsar JD Jr, Eddie D, Walter J. A randomized trial comparing the Tennant Biomodulator to transcutaneous electrical nerve stimulation and traditional Chinese acupuncture for the treatment of chronic pain in military service members. Mil Med Res. 2019 Dec 2;6(1):37. doi: 10.1186/s40779-019-0227-4. PMID 31791416